CLINICAL TRIAL: NCT03107923
Title: Better Patient Selection to Transcatheter Aortic Valve Implantation
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Per Steinar Halvorsen, Consultant and research group leader, Oslo University Hospital
Other Study IDs: 535444
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Aortic Valve Stenosis; Left Ventricular Dysfunction; Myocardial Fibrosis
Keywords: Myocardial fibrosis; Aortic Valve Stenosis; TAVI; Outcome
MeSH Terms: conditions — Aortic Valve Stenosis; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Routine blood tests on admittance and after one year. These include markers of heart failure as S-proBNP/troponin and kindey failure as S-kreatinin/S-Cystatin C, electrolytes, Hgb
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preoperative myocardial reserve yes/no: Patients with extensive myocardial fibrosis typically presents with limited myocardial contractile reserve that can be assessed by a dobutamine stress test. The patients will be allocated to a responder and non-responder group according to the results from this test.
  Interventions: Diagnostic Test: Dobutamine stress test

INTERVENTIONS:
Diagnostic Test: Dobutamine stress test — Test of myocardial reserve

SUMMARY:
This study evaluates whether a preoperative assessment of myocardial contractile reserve by tissue Doppler Imaging and myocardial fibrosis by cardiac magnetic resonance imaging (MRI) can enhance the patient selection and risk stratification to transcatheter aortic valve implantation.

DETAILED DESCRIPTION:
In this prospective observation study we will investigate whether a preoperative test of myocardial contractile reserve can predict adverse outcome after TAVI. We intend to examine preoperative myocardial contractile reserve by use a low dose dobutamine test and relate this to pre-existing myocardial focal and diffuse myocardial fibrosis detected by new cardiac magnetic resonance imaging (MRI) methods and new echocardiographic methods. These measures will be primarily related to long term (12 months) mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients declined surgical aortic valve replacement and scheduled for transfemoral aortic valve implantation.

Exclusion Criteria:

* Aortic valve endocarditis
* aortic annulus >31mm
* preoperative pacemaker
* severe aortic insufficiency (>grad 3)
* rapid atrial fibrillation
* unprotected left main coronary stenosis not suitable for percutaneous intervention.
* unstable angina
* life expectancy less than 12 months
* mental disorder including dementia and condition which interferes with protocol compliance.
* renal failure (glomerular filtration rate < 45 ml/min/m2), only have T1 mapping by CMRI.
* Patients with metal not suitable for MRI.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for transfemoral aortic valve implantation at Oslo University Hospital-Rikshospitalet
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
MACE | 1 year
  MACE at 12 months follow-up after TAVI, MACE definition: rehospitalization for heart failure or other valve related complications, nonfatal myocardial infarction, nonfatal stroke, or (cardiovascular) death

SECONDARY OUTCOMES:
NYHA functional classification of heart failure, Lack of improvement and/ or function class III or IV 12 months after the procedure defined unfavorable outcome | 1 year
  Number of Participants hospitalizated for heart related diseases during 12 month follow-up.
Patient quality of life (QoL) | 1 year
  Quality of life record (SF 36), Physical function (age adjusted normal value 71.6 (SD 26.9)) and Physical role (age adjusted normal value 57.0 (SD 43.8)) , the patients were divided into groups using the predefined minimal change of 15 and 18,75 points, respectively. Changes above these tresholds at 12 month follow-up indicat better QoL outcomes.
6 Minute Walking Test | 1 year
  Favorable outcome defined as improvement in walking distance of 30 meters or longer at one year follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Fosse, Professor, Study Director — The Intervention Centre, Oslo University Hospital
Locations (2):
- Norway (2):
  - Oslo Universtity Hospital, Oslo
  - The Intervention Centre, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bax JJ, Delgado V, Bapat V, Baumgartner H, Collet JP, Erbel R, Hamm C, Kappetein AP, Leipsic J, Leon MB, MacCarthy P, Piazza N, Pibarot P, Roberts WC, Rodes-Cabau J, Serruys PW, Thomas M, Vahanian A, Webb J, Zamorano JL, Windecker S. Open issues in transcatheter aortic valve implantation. Part 1: patient selection and treatment strategy for transcatheter aortic valve implantation. Eur Heart J. 2014 Oct 7;35(38):2627-38. doi: 10.1093/eurheartj/ehu256. Epub 2014 Jul 25. PMID 25062952
- [Background] Eidet J, Dahle G, Bugge JF, Bendz B, Rein KA, Aaberge L, Offstad JT, Fosse E, Aakhus S, Halvorsen PS. Long-term outcomes after transcatheter aortic valve implantation: the impact of intraoperative tissue Doppler echocardiography. Interact Cardiovasc Thorac Surg. 2016 Sep;23(3):403-9. doi: 10.1093/icvts/ivw159. Epub 2016 May 30. PMID 27241050
- [Derived] Saevik M, Andersen MH, Beitnes JO, Aaberge L, Halvorsen PS. Health Related Quality of Life (HRQoL) after transcatheter aortic valve implantation in aortic stenosis patients: exploring a novel threshold for clinically significant improvement after 12 months. J Patient Rep Outcomes. 2025 May 26;9(1):58. doi: 10.1186/s41687-025-00894-1. PMID 40418351